CLINICAL TRIAL: NCT00366366
Title: Phase III, Open, Randomised Immunogenicity and Reactogenicity Study to Assess the Interchangeability Between GSK Bios' DTPa-HBV-IPV/Hib and DTPa-IPV/Hib + HBV at 3rd Dose of Primary Vac. Course in Children Who Received HBV Vac. at Birth and One Month of Age and DTPa-IPV/Hib Vac at 3-4 Mth of Age
Brief Title: To Evaluate Immunogenicity & Safety of GSK Bio's DTPa-HBV-IPV/Hib (Mixed Vaccine) and DTPa-IPV/Hib + HBV Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217744/075
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

INTERVENTIONS:
Biological: Infanrix-Hexa

SUMMARY:
This study assessed the immunogenicity and safety of two vaccination regimens that employed either GSK Biologicals' combined DTPa-HBV-IPV/Hib vaccine or DTPa-IPV/Hib vaccine. In the two groups, infants received the DTPa-IPV/Hib vaccine at 3 and 4 months of age, as the first 2 doses of the primary vaccination course. At 5 months of age, they received either the DTPa-IPV/Hib vaccine co-administered with the HBV vaccine or a dose of the DTPa-HBV-IPV/Hib vaccine as a 3rd dose. Infants in the two groups had previously received 2 doses of HBV vaccine at birth and at 1 month of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant at the age of 11 - 17 weeks.
* Written informed consent obtained from the parents or guardians of the subject.
* Free of obvious health problems as established by clinical examination before entering into the study.
* Hepatitis B vaccine at birth and one month of age.

Exclusion Criteria:

* Previous vaccination against measles, mumps, rubella and/or varicella.
* Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* A family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection.
* Major congenital defects.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.

Ages: 11 Weeks to 17 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2001-09; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Anti-HBs conc >=10 mIU/ml, 1 month after the last vaccine dose

SECONDARY OUTCOMES:
Ab conc/titers against all vaccine antigens
Safety: Solicited symptoms, unsolicited AEs and SAEs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lim FS, Han HH, Jacquet JM, Bock HL. Primary vaccination of infants against hepatitis B can be completed using a combined hexavalent diphtheria-tetanus-acellular pertussis-hepatitis B-inactivated poliomyelitis-Haemophilus influenzae type B vaccine. Ann Acad Med Singap. 2007 Oct;36(10):801-6. PMID 17987229
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 217744/075 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 217744/075 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 217744/075 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 217744/075 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 217744/075 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 217744/075 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register